CLINICAL TRIAL: NCT03922958
Title: Immunoparalysis in Acute Kidney Injury After Cardiac Surgery
Status: Terminated | Type: Observational
Why Stopped: funding ended
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0127
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury; Immune Deficiency
MeSH Terms: conditions — Acute Kidney Injury; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples and urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infection and sepsis are common after acute kidney injury (AKI) and increase mortality. In this study, the investigators will determine whether patients with acute kidney injury after cardiac surgery have immunosuppression as judged by blood markers of immunoparalysis.

DETAILED DESCRIPTION:
Immunoparalysis is an immunosuppressed state that occurs after a wide variety of insults including sepsis and cardiopulmonary bypass surgery. Due to the impaired infection fighting ability, patients with immunoparalysis are at risk of subsequent infection which can increase mortality. Immunoparalysis can be measured by two methods: 1) ex vivo endotoxin stimulation and 2) blood monocyte HLA-DR levels. Since sepsis is also a known complication of Acute Kidney Injury(AKI), the investigators hypothesize that AKI is a risk factor for immunoparalysis. The investigators plan to look at these blood factors of immune function from patients before and 3 days following cardiac surgery. Urine will also be collected from the patients before their surgery as well as the 3 days following for AKI biomarker measurement. This prospective cohort will enroll 300 patients and determine the duration and severity of immunoparalysis among patients who develop AKI and those who do not develop AKI.

ELIGIBILITY:
Inclusion Criteria:

* All adults undergoing cardiac surgery with CPB will be considered for enrollment.

Exclusion Criteria:

* Factors that affect immune function or AKI assessment are the basis for exclusion criteria:

  * Concurrent disease associated with immunosuppression including malignancy, chronic infection (e.g., HIV, Hepatitis C), organ transplant and immunosuppressant medications
  * Documented acute infection with the past 1 month (e.g., pneumonia, urinary tract infection)
  * Prednisone or other steroid use currently or within the past one month
  * AKI at the time of surgery
  * ESRD requiring renal replacement therapy
  * Estimated GFR <45 mL/min (as judged by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing cardiac surggery with CPB at University of Colorado Hospital (UCH)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Determine if patients with AKI have a higher rate of immunoparalyisis after CPB | 2 years
  Patients with AKI will have a higher rate of immunoparalysis compared to those without AKI when immunoparalysis is identified by TNF levels after ex vivo endotoxin stimulation. As well as patients with AKI will have a higher rate of immunoparalysis compared to those without AKI when immunoparalysis is identified by monocyte HLA-DR (mHLA-DR) expression.
Determine if the severity of immunoparalysis is greater among patients with AKI after CPB compared to patients without AKI after CPB. | 2 years
  Patients with more severe AKI (based on KDIGO stage) will have a greater severity of immunoparalysis based on lower TNF levels after ex vivo endotoxin stimulation or lower mHLA-DR. As well as among the entire cohort, a greater increase in serum creatinine from baseline will be associated lower TNF levels after ex vivo endotoxin stimulation or lower mHLA-DR.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Faubel, MD, Principal Investigator — UC Denver Anschutz Medical Campus
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States